CLINICAL TRIAL: NCT04857593
Title: Online Singing Interventions for Postnatal Depression in Times of Social Isolation: a Single Arm Study
Acronym: SHAPER-PNDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 219425/Z/19/Z-PNDO
Record Dates: First submitted 2021-03-18; First posted 2021-04-23 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-02

CONDITIONS: Postnatal Depression; Social Isolation
Keywords: singing; depression; music; social isolation; anxiety; postnatal; mental health; perinatal
MeSH Terms: conditions — Depression, Postpartum; Social Isolation; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): M4M online is a 6-week intervention for mothers with PND. The original M4M programme would be delivered face-to-face in groups of 8-12 mothers in weekly sessions lasting one hour. However, due to the current situation with COVID-19, we will therefore modify the original face-to-face intervention for this online study, as follows:
  * Run groups of around 15-17 women to ensure that all participants can be visible on one screen during online delivery to create a stronger sense of community and connection
  * Offer 6 weeks of intervention, also building on the evidence from the face-to-face intervention that by 6 weeks there is already a significant improvement in depressive symptoms compared with control interventions24
  * Introduce a two-week lead-in period before the beginning of the six-session course, where mothers will be able to use WhatsApp and at least one (monitored) Zoom session to get to know each other.
  Interventions: Behavioral: Melodies for Mums

INTERVENTIONS:
Behavioral: Melodies for Mums — Classes start with a chat between mothers and the artist. The singing session will include welcome songs, introducing the babies and mothers to one another, and then involve a range of singing and music activities. These will include learning songs from around the world, ranging from short vocal exercises that use "motherese" style noises and sound effects (including sound baths where the mothers sang a sustained note providing a relaxation technique), to simple lullabies that can be picked up very quickly and sung in basic harmonies or rounds, to longer or more complex songs that will be learnt gradually over the weeks. Instruments such as guitar and ukulele will also be used by the artist for a small number of songs. Mothers will also work to write some of their own songs over the weeks, developing lyrics together about their babies or experiences of motherhood and creating simple melodies. Classes will be led by workshop leaders trained by Breathe, with support of assistants.

SUMMARY:
Melodies for Mums (M4M) is an intervention developed and tested as part of a collaboration between the Royal College of Music, Imperial College London and University College London from 2015-2017. The programme involved weekly singing classes for mothers and babies delivered in groups of 8-12 participants in Children's Centres for 10 weeks. M4M was tested in a three-arm RCT involving 134 mothers with PND (with an Edinburgh Postnatal Depression Scale (EPDS) score above 10), compared with a comparison group (10 weeks of creative play classes) or care as usual (wait-list control). The study found that mothers with moderate-severe symptoms of PND who participated in the programme with their baby had a significantly faster improvement in symptoms than mothers in usual care. Specifically, the mothers in the singing group had an average EPDS score of 15.7 at baseline (moderate depression), which dropped to 10.3 by week 6 and 9.4 by week 10. This improvement equated to an average 35% decrease in depressive symptoms across the first 6 weeks, by which point 65% of the singing group no longer had an EPDS above 13.

While funding has been secured to upscale this intervention as part of the SHAPER-PND programme, funded by the Wellcome Trust, the recent lockdown has not only halted the programme in its face-to-face format, but also prompted the interest in developing an online version that can be used (1) if the requirement for social distancing, even when the lockdown is relaxed, makes impossible the delivery of the programme; and (2) to broaden the reach to a nationwide delivery and extending to a wider population that may not have been able to attend in-person sessions due to geographical constraints or severity of symptoms.

M4M online is a 6-week intervention for mothers with PND. The original M4M programme would be delivered face-to-face in groups of 8-12 mothers in weekly sessions lasting one hour. However, due to the current situation with COVID-19, we will therefore modify the original face-to-face intervention for this online study, as follows:

* Groups of around 15-17 women to ensure that all participants can be visible on one screen during online delivery to create a stronger community and connection
* Offer 6 weeks of intervention, also building on the evidence from the face-to-face intervention that by 6 weeks there is already a significant improvement in depressive symptoms compared with control interventions
* Introduce a two-week lead-in period before the beginning of the six-session course, where mothers will be able to use WhatsApp and at least one (monitored) Zoom session to get to know each other.

DETAILED DESCRIPTION:
This single-arm clinical trial aims, in a period of 12 months, to pilot and evaluate an online delivery of Melodies for Mums with the ambition:

1. To develop a remote intervention that can become a mainstream therapeutic tool not only at times of social isolation and distancing, but also for mothers who cannot leave their houses (e.g. because of mental health difficulties or medical comorbidities) or who live in areas where the intervention is unavailable;
2. To create a separate control group to the original face-to-face intervention, as the investigators are still aiming to deliver the original SHAPER-PND when the investigators will be able to start again; and
3. To make the best use of the expertise/experience available within the researchers and artists community brought together by the Wellcome Trust funding for the SHAPER-PND study.

In light of the limitations imposed by the current pandemic, the investigators aim to deliver M4M using a virtual platform to replace the in-person singing sessions. To achieve this, the investigators will deliver a more advanced version of a 'virtual choir' but keeping to the framework of the existing M4M programme; the investigators take the learnings by Breathe Arts Health Research from their Breathe Sing group for individuals with respiratory conditions. Prior to lockdown, this group met fortnightly in-person to use singing to benefit physical and mental health. During the COVID-19 pandemic, this group has moved online and is continuing to have excellent uptake with weekly attendance numbers higher than when the group was delivered in-person. M4M online will take a similar format, consisting of weekly sessions of one hour each, where women connect via Zoom and sing from their home while following the leader. To avoid the inevitable problems with Wi-Fi delays and instability, all participants are muted at certain times in the session but can all hear the singing leader throughout. The singing leader will also use a backing track that will be recorded specifically to support delivery, and has other voices and harmonies included to amplify the experience of singing with others. An additional Breathe member of staff will support participants to set up the online connection before the sessions and help them troubleshoot during the session. All participants are also connected via a WhatsApp group (monitored by Breathe), and there will be a space at the beginning and end of the sessions where all participants are unmuted and can chat with the artist or their peers, in an unstructured way.

M4M online will be delivered as a single-arm clinical trial, without a control group. Participants will be recruited in the community, mostly via social media and other signposting methods according to the usual procedures carried out by Breathe for recruiting into the face-to-face M4M programme but with enhanced advertisement and social media reach nationally. Before entering the study, mothers will be assessed by the research team, and if eligible, will be allocated to a singing group for 6 weekly sessions. Participants will remain in the same group to allow greater sense of community and familiarity with the artist, facilitator, and the other participants. Participants will be regularly assessed by the researchers and if they give consent, will provide biological samples. Follow up will be carried out 10 and 26 weeks after completion of the trial.

Setting: This is a single-centre trial that will be run online across the UK via the platform Zoom. In order to enrol a sufficiently large sample of women, there will be 4 blocks of the 6-week singing sessions in total. Women will be followed up at weeks 16 and 32.

Recruitment will be primarily done through:

* Posters and flyers in baby weigh clinics and other community and clinical centres for postnatal mothers and their babies, if lockdown rules allow that;
* Signposting via other health and social care professionals and in the community via email contacts;
* Social media/online forums
* Self-referral following general advertisement Community services will be made aware of the study through a poster/flyer/e-mail campaign sent directly to them. Breathe has a database of contacts used to recruit for Breathe's Melodies for Mums in-person programme that will be used for this purpose.

In terms of social media recruitment, the following will be used: various Facebook targeted groups, Instagram & Twitter hashtags to find groups and forums to promote to, plus more traditional routes e.g. to get local authorities to advertise as part of their various tiers of information of available local services.

The first contact will be done by Breathe Arts staff over the phone, following social media/online self-referral/direct self-referral through posters/flyers in community and clinical centres. The research team will only become involved once the potential participants have made contact with the Breathe Arts team, completed an online screening form and given consent for the basic information collected onto the online screening (personal information, EPDS score) to be shared with the research team.

All potential participants will initially be directed to a pre-screening online form on Breathe's website. This will capture basic information including the mother's name, date of birth (DOB), baby's DOB, address, telephone number, and once this has been submitted, they will be sent EPDS scale to complete. Women will be asked to read an online participant information sheet (PIS) and to electronically confirm consent after reading the informed consent form (ICF) to their personal data being collected. The PIS will explain that their details will be used for further contact related to the trial in case their EPDS score is equal or higher than 10.

If a woman's EPDS score is lower than 10, she will receive a notification that she is not currently eligible to participate and will receive information on other support services in the meantime. In the consent form, it will be asked if she would like to be re-contacted at a future date when the next series of workshops is scheduled, and if she agrees, she will be contacted in the same way as other women who express interest for the first time and screened again. Researchers will wait at least 1 month before inviting re-screening.

If a woman's score is 10 or higher, she will be notified that she is potentially eligible and when a new round of 6 singing sessions becomes available, the research team will arrange a call to undertake the full screening interview against the inclusion/exclusion criteria. This full screening will take place in the 2 full weeks prior to the online classes starting (referred to as 'Baseline'). If the participant is found to be non-eligible, they will be given information for other support services. If the participant is found to be eligible the researcher will carry out the baseline measures. A contact point will be made available for participants in case they wish to ask further questions regarding the trial. If more women are found to be eligible for each 6-week programme than the sessions have capacity for, then priority will be given to those with the highest EPDS scores. The others will be invited to rescreen for the next group.

A copy of the ICF will be sent electronically to the participant once the baseline Zoom call has been arranged. The ICF will include a section detailing the samples to be collected (saliva) and others measures to be analysed, as well as the consent to obtain babies' data (in video and other formats) and babies' saliva samples throughout the study (see full table for more information on measures in section 9.7). A participant can opt out of the sample collections or babies' data collection and enter the trial for all other measures. The Informed consent will also include a point stating that the participants might be contacted for further studies. This will allow for the sample of the population enrolled on the trial to be approached for future follow-up research questions.

Recruitment of deliverers:

During the course of the study, deliverers will be recruited by the research team from the pool of 1-3 artists trained by Breathe that deliver the M4M sessions. Researchers will approach deliverers to ascertain their interest level in participating in our study. Deliverers will be recruited for the purpose of assessing the ways in which this 6-week online singing programme can ameliorate mothers' postnatal depression.

If deliverers express interest, researchers will provide them with the Deliverer participant information sheet, which will explain to them why the researchers are interested in incorporating deliverer feedback on the programme into our study, and will explain what kind of information the researchers are looking to collect from them. The researchers will then electronically provide deliverers who are interested with the deliverer informed consent form to consent to their personal data being collected.

The ICF will explain that data will be collected and stored confidentially, and will have the option to opt-in to each consent point.

If deliverers consent, the UCL researcher will arrange a Zoom call with them, during which the researchers will interview them and collect feedback on how they felt the programme helped women's postnatal depression, with the aim to use their views/experiences to help inform upon the development of the programme.

Safeguarding

The research teams will have three safeguarding check points:

1. The UCL research team will check the EPDS scores of all participants as they come through online (baseline, 3, 6, 16 and 32 weeks) at least once a week, and they will alert the clinical leads of the study if (a) EPDS scores are more than 25 out of 30 or, (b) EPDS includes a score of 2 or more on the self-harm question.
2. Breathe will report to the KCL research team on any concerns during intervention sessions within 24 hours of noting the concern, especially if the behaviour is felt to be indicative that they are at immediate risk of harming themselves or their babies.
3. If the research team thinks that the behaviour (or any responses to the questionnaires collected) of any participant during the online assessments or during any other contact (e.g. phone contact), is felt to be indicative that they are at immediate risk of harming themselves or their babies or others, the same process will be taken.

The clinical leads (the perinatal psychiatrists) on the research team will assess each report and decide whether there is a need to contact a participant, alert a participant's GP or contact any other healthcare services. This decision will be made within 72 hours of receiving the report. Participants will be informed of this process in the PIS. If contact with a health professional is being made on behalf of a participant, the participant will be informed that this is taking place.

Assessments Participants will be assessed via Zoom for baseline, week 6 and week 32 assessments. Week 3 and 16 assessments will be completed online by the mothers only, due to the self-reporting nature of the measures. It is expected that all mothers will have access to an internet-enabled device, as this is an essential inclusion criterion. For baseline online measures, participants will be encouraged to complete these a day either side of the first session. For week 3 measures, participants will be encouraged to complete these within 3 days of the session. However, in order to allow flexibility in the schedule, a +/-1 week variation in the date of collection of the measures will be accepted (apart from week 6, when the window will be weeks 6-8).

Individual qualitative interviews with a sub sample of women will take place after the final session of the intervention either by telephone or video call. Interviews will also be conducted with the intervention deliverers/singing group leaders, the deliverers. The interviews will explore the experiences, mechanisms of effect, barriers and facilitators to taking part and delivering online singing groups.

Sample collection and transportation Participants can opt out of sample collection at any stage of the study. Samples will be labelled according to participant ID allocated at randomisation so that the samples will not be directly linked to any personal data.

All saliva samples will be collected by Salivette absorbent swabs for adults and SalivaBio Children's Swabs for babies and used to measure cortisol levels. Mothers will be asked to collect samples to measure diurnal cortisol rhythm and cortisol reactivity to the sessions.

For diurnal samples, mothers will be asked to collect six saliva samples from themselves (awakening, +15, +30+ and +60 min after awakening, at 12 noon and 8 pm), and two samples from their baby (awakening and 8pm). Mothers will be asked to collect these samples up to 3 days prior to their session (baseline, week 3 and week 6), however, in order to allow flexibility in the schedule, a +/-5 day variation will be accepted in the date of collection. The investigators have extensively experience with this methodology and successfully collected such data before.

Mothers will also be asked to collect saliva samples from themselves and their baby immediately before and after their session (week 1, week 3 and week 6).

Mothers will be provided with pre-paid envelopes in which to return both diurnal and session samples together for each time point. All samples should be kept in the mother's fridge until ready to return by post.

Follow-up data collection Upon termination of the 6 weekly sessions, participants will be contacted to complete follow-up questionnaires around weeks 16 and 32. An additional virtual assessment will be carried out around week 32. A sub sample of women will be invited to take part in a qualitative interview about their experiences of receiving the online intervention up to two weeks after their final intervention session.

ELIGIBILITY:
Inclusion Criteria

* Women aged 18 or older
* Satisfactory understanding of English
* Women who have a child between 0 and up to 9 months old
* Women with postnatal depression diagnosed using symptoms of PND at a minimum score of 10 on the EPDS.

Exclusion Criteria

The participant may not enter the study if ANY of the following apply:

* Child outside of the age-range specified
* Unable to give informed consent
* Unable

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmine M Pariante, Principal Investigator — King's College London - IoPPN
Locations (1):
- Maurice Wohl Clinical Neuroscience Institute, 5 Cutcombe Rd, Brixton, London SE5 9RT, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 12 months and ending 36 months following article publication.
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Background] Fancourt D, Perkins R. Effect of singing interventions on symptoms of postnatal depression: three-arm randomised controlled trial. Br J Psychiatry. 2018 Feb;212(2):119-121. doi: 10.1192/bjp.2017.29. PMID 29436333
- [Background] Green P. Risks to children and young people during covid-19 pandemic. BMJ. 2020 Apr 28;369:m1669. doi: 10.1136/bmj.m1669. No abstract available. PMID 32345583
- [Background] Fancourt D, Steptoe A. Present in Body or Just in Mind: Differences in Social Presence and Emotion Regulation in Live vs. Virtual Singing Experiences. Front Psychol. 2019 Apr 10;10:778. doi: 10.3389/fpsyg.2019.00778. eCollection 2019. PMID 31024405
- [Derived] Bind RH, Sawyer K, Hazelgrove K, Rebecchini L, Miller C, Ahmed S, Dazzan P, Sevdalis N, Bakolis I, Davis R, Lopez MB, Woods A, Crane N, Manoharan M, Burton A, Dye H, Osborn T, Greenwood L, Perkins R, Fancourt D, Pariante CM, Estevao C. Feasibility, clinical efficacy, and well-being outcomes of an online singing intervention for postnatal depression in the UK: SHAPER-PNDO, a single-arm clinical trial. Pilot Feasibility Stud. 2023 Jul 27;9(1):131. doi: 10.1186/s40814-023-01360-9. PMID 37501172
- [Derived] Bind RH, Estevao C, Fancourt D, Hazelgrove K, Sawyer K, Rebecchini L, Miller C, Dazzan P, Sevdalis N, Woods A, Crane N, Manoharan M, Burton A, Dye H, Osborn T, Greenwood L, Bakolis I, Lopez MB, Davis R, Perkins R, Pariante CM. Online singing interventions for postnatal depression in times of social isolation: a feasibility study protocol for the SHAPER-PNDO single-arm trial. Pilot Feasibility Stud. 2022 Jul 18;8(1):148. doi: 10.1186/s40814-022-01112-1. PMID 35851430

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: M4M online is a 6-week intervention for mothers with PND.
  * Offer 6 weeks of intervention, also building on the evidence from the face-to-face intervention that by 6 weeks there is already a significant improvement in depressive symptoms compared with control interventions24
  * Introduce a two-week lead-in period before the beginning of the six-session course, where mothers will be able to use WhatsApp and at least one (monitored) Zoom session to get to know each other.
  Melodies for Mums: Classes start with a chat between mothers and the artist. The singing session will include welcome songs, introducing the babies and mothers to one another, and then involve a range of singing and music activities. These will include learning songs from around the world, ranging from short vocal exercises that use "motherese" style noises and sound effects (including sound baths where the mothers sang a sustained note providing a relaxation technique), to simple lullabies that can be picked up very quickly and sung in basic harmonies or rounds, to longer or more complex songs that will be learnt gradually over the weeks. Instruments such as guitar and ukulele will also be used by the artist for a small number of songs. Mothers will also work to write some of their own songs over the weeks, developing lyrics together about their babies or experiences of motherhood and creating simple melodies. Classes will be led by workshop leaders trained by Breathe, with support of assistants.
Period: Overall Study
Arm/Group | Intervention
Started | 37
Completed | 32
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: New mothers with postnatal depression
Groups:
- M4M Intervention: We modified the original face-to-face intervention for this online study as follows:
  Groups were up to 15 women (in line with the community M4M) to ensure all participants were visible on one screen and thus create a stronger sense of community and connection.
  The intervention was 6 weeks long, based on the face-to-face intervention evidence that by 6 weeks, there is already a significant improvement in depressive symptoms compared with control interventions.
  Mothers were connected from week 2 of the intervention to an optional WhatsApp group, to mirror the social interaction component of the in-person community intervention.
  Artists were trained centrally by Breathe to ensure that fidelity to the original M4M was maintained. Furthermore, a member of Breathe was present on each Zoom singing session to monitor and ensure the session was being delivered according to protocol. During the singing portion of the sessions, all participants were muted, while the artist was unmuted and playing background melodies, to ensure a group feeling while avoiding broadband-related sound delays and other background noises. Thus, participants could hear themselves, the artist, and the background melody, with pre-recorded voices, that recreated the community M4M setting. Outside of sessions, mothers had access to a weblink with M4M songs, to allow them to sing at home in between sessions and beyond M4M.
Arm/Group | M4M Intervention
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.3 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Maternal Ethnicity: White | 28
  Maternal Ethnicity: Ethnic minority groups | 9
Region of Enrollment [Number; unit: participants]
  United Kingdom | 37
Marital Status [Count of Participants; unit: Participants]
  Married/cohabiting | 34
  Single with/without partner | 3
Biological Father Ethnicity [Count of Participants; unit: Participants] — Not collected from one participant. Population: Number of participants we obtained measure from
  Participants
    number analyzed (Participants) | 36
    White | 26
    Ethnic minority groups | 10
Maternal Qualifications [Count of Participants; unit: Participants]
  Higher education or above | 33
  GCSE/A-level or below | 4
Maternal Employment Status [Count of Participants; unit: Participants]
  Employed/student/maternity leave | 32
  Unemployed/full-time mother | 5
Partner Employment Status [Count of Participants; unit: Participants]
  Employed/student | 35
  Missing | 2
Household income [Count of Participants; unit: Participants]
  Less than £30,000 | 2
  £30,000 or greater | 35
Infant Age [Mean (Standard Deviation); unit: Months] | 4 (2.5)
Infant Sex [Count of Participants; unit: Participants]
  Female | 18
  Male | 19
Attending Other Mother-Baby Groups [Count of Participants; unit: Participants]
  Yes | 17
  No | 20
Childhood Experience of Abuse [Count of Participants; unit: Participants] — Not collected from four participants. Population: Number of participants we obtained measure from
  Participants
    number analyzed (Participants) | 33
    Yes | 12
    No | 21
Adult Experience of Intimate Partner Violence [Count of Participants; unit: Participants]
  Yes | 15
  No | 22
Intrusive Life Event Across Lifetime [Count of Participants; unit: Participants] — Not collected from four participants. Population: Number of participants we obtained measure from
  Participants
    number analyzed (Participants) | 33
    Yes | 16
    No | 17
Threatening Life Event in Perinatal Period [Count of Participants; unit: Participants] — Not collected from four participants. Population: Number of participants we obtained measure from
  Participants
    number analyzed (Participants) | 33
    Yes | 18
    No | 15
Current Diagnosis of MDD [Count of Participants; unit: Participants]
  Yes | 22
  No | 15
Lifetime Diagnosis of MDD [Count of Participants; unit: Participants]
  Yes | 28
  No | 9

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Effectiveness of Online Group Singing Interventions on Symptoms of Postnatal Depression Using the Edinburgh Postnatal Depression Scale (EPDS)
Description: To assess the effectiveness of online group singing interventions on symptoms of postnatal depression using the Edinburgh Postnatal Depression Scale (EPDS)
  The EPDS was developed to assist health professionals in detecting mothers suffering from Postnatal depression. The scale consists of 10 short statements. A mother checks off one of four possible answers that is closest to how she has felt during the past week. The EPDS is measured on a scale of 0-30, where a higher score indicates more severe depression. Mothers scoring above 12 or 13 are likely to be suffering from depression.
Time Frame: The primary outcome measure is changes in EPDS total score between baseline and Week 6 (end of treatment).
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Singing group: This is a single-arm trial in which all participants are allocated to our online Melodies for Mums singing intervention.
Arm/Group | Singing group
Number analyzed (Participants) | 37
score on a scale
  Mean EPDS score at baseline | 16.6 (3.7)
  Mean EPDS score at week 6 | 11.2 (5.3)
Statistical Analysis 1: Comparison: Singing group; Test type: Other; p = .001, t-test, 2 sided; Mean change in EPDS score = 5.4

2. Secondary Outcome: To Assess Whether Online Singing Improves (Changes) Further Aspects of Mental Health, Including Depression Using the Hamilton Depression Rating Scale (HDRS)
Description: To assess whether online singing improves (changes) further aspects of mental health, including depression, using:
  Hamilton Depression Rating Scale (HDRS): is a semi-structured clinician-administered depression assessment scale. Scoring is from 0-52 and is based on the 17-item scale, where each question receives a score from either 0-2 or 0-4, depending on the question. Total summed scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score being 52 on the 17-point scale.
Time Frame: Compare changes between baseline and weeks 6 (end of treatment).
Population: Single-arm group who participated in online Melodies for Mums intervention
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Singing group: Change in Hamilton Depression Rating Scale score between baseline and end of intervention
Arm/Group | Singing group
Number analyzed (Participants) | 37
units on a scale
  Baseline | 13.8 (6.3)
  Week 6 | 7.4 (6.8)

3. Secondary Outcome: To Assess Whether Online Singing Improves (Changes) Further Aspects of Mental Health, Including Depression Using the Beck Depression Inventory (BDI).
Description: To assess whether online singing improves (changes) further aspects of mental health, including depression, using:
  Beck Depression Inventory (BDI): is a 21-item, self-rated scale that evaluates key symptoms of depression. Total scores range from 0-63. Each item is rated 0-3, whereby a higher score indicates more severe depression. Scores from each question are summed to calculate the total score. 1-10 is considered normal; 11-16 is mild mood disturbance; 17-20 is borderline clinical depression; 21-30 is moderate depression; 31-40 is severe depression; 40 and above is extreme depression.
Time Frame: Compare changes between baseline and weeks 3, 6, 16, 32.
Population: Change in Beck Depression Inventory score across entire study period (baseline, week 3, week 6, week 16, week 32) in single-arm group who received online Melodies for Mums singing intervention.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Singing group: Change in Beck Depression Inventory score across entire study period (baseline, week 3, week 6, week 16, week 32) in single-arm group who received online Melodies for Mums singing intervention.
Arm/Group | Singing group
Number analyzed (Participants) | 37
score on a scale
  Baseline | 18.9 (6.6)
  week 3 | 15.1 (7.5)
  week 6 | 13.0 (8.6)
  week 16 | 12.3 (8.4)
  week 32 | 11.6 (8.1)

4. Secondary Outcome: To Assess Whether Online Singing Improves (Changes) Further Aspects of Mental Health, Including Stress Using the Perceived Stress Scale (PSS)
Description: To assess whether online singing improves (changes) further aspects of mental health, including stress.
  Stress will be evaluated using the following scale:
  Perceived Stress Scale (PSS): is an 10-item questionnaire assessing one's perceived stress levels. Each question is scored 0-4 and totals from each question are summed to calculate total score, which can range from 0-40. Each question must be answered on a likert scale, ranging from 'never' (0) to 'very often', (4), whereby a higher score indicates greater stress.
Time Frame: Compare changes between baseline and weeks 3, 6, 16, 32.
Population: Change in Perceived Stress Scale score across entire study period (baseline, week 3, week 6, week 16, week 32) in single-arm group who received online Melodies for Mums singing intervention.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Singing group: Change in Perceived Stress Scale score across entire study period (baseline, week 3, week 6, week 16, week 32) in single-arm group who received online Melodies for Mums singing intervention.
Arm/Group | Singing group
Number analyzed (Participants) | 37
score on a scale
  Baseline | 29.0 (5.7)
  Week 3 | 22.4 (5.2)
  Week 6 | 19.7 (5.3)
  Week 16 | 19.2 (5.7)
  Week 32 | 19.1 (6.1)

5. Secondary Outcome: To Assess Whether Online Singing Improves (Changes) Further Aspects of Mental Health, Including Wellbeing Using the Office for National Statistics Wellbeing Scale (ONS):
Description: Wellbeing will be evaluated using the following scale:
  Office for National Statistics Wellbeing Scale (ONS): is a four-item questionnaire assessing life satisfaction, worthwhile, happiness, and anxiety. People are asked to respond to the questions on a scale from 0 to 100 where for life satisfaction/worthwhile/happiness a higher score indicates greater wellbeing, and for anxiety a greater score indicates greater anxiety. Total scores can range from 0-100.
Time Frame: Compare changes between baseline and weeks 3, 6, 16, 32.
Population: Change in Office for National Statistics Wellbeing Scale score between baseline and end of intervention
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Singing group: Change in Office for National Statistics Wellbeing Scale score between baseline and end of intervention
Arm/Group | Singing group
Number analyzed (Participants) | 37
score on a scale
  Baseline life satisfaction | 50.0 (23.0)
  Week 6 life satisfaction | 72.8 (11.7)
  Baseline worthwhileness | 51.7 (34.0)
  Week 6 worthwhileness | 78.6 (15.1)

6. Secondary Outcome: To Assess Whether Online Singing Improves (Changes) Further Aspects of Mental Health, Including Anxiety, Using the State-Trait Anxiety Scale (STAI)
Description: Anxiety will be evaluated using the following scale:
  State-Trait Anxiety Scale (STAI): is a self-rated questionnaire which assesses intensity or frequency of anxiety. It is divided into two sections, one measuring 'state' and the other 'trait' of anxiety. We have analysed the 'state' section of the STAI (STAI-S). The STAI-S consists of 20 questions, which can be scored from 1-4 and then summed. The range of possible scores is 20 to 80, whereby a higher score indicates greater anxiety. A cut-off score of at least 40 has been considered to be clinically meaningful.
Time Frame: Compare changes between baseline and weeks 3, 6, 16, 32.
Population: Change in State Trait Anxiety Inventory score across entire study period (baseline, week 3, week 6, week 16, week 32) in single-arm group who received online Melodies for Mums singing intervention.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Singing group: Change in State Trait Anxiety Inventory score across entire study period (baseline, week 3, week 6, week 16, week 32) in single-arm group who received online Melodies for Mums singing intervention.
Arm/Group | Singing group
Number analyzed (Participants) | 37
score on a scale
  Baseline | 48.4 (27.1)
  Week 3 | 41.7 (26.8)
  Week 6 | 37.1 (26.8)
  Week 16 | 37.9 (26.7)
  Week 32 | 37.2 (25.9)

7. Secondary Outcome: To Ascertain Whether Online Singing Improves the Observed Mother-infant Interaction Using the Crittenden CARE-Index (CCI)
Description: To assess whether the online singing intervention improves upon aspects of the mother-infant relationship.
  The observed mother-infant interaction will be assessed using:
  Crittenden CARE-Index (CCI): The CCI is a validated tool to clinically assess the mother-infant interaction. Videos are filmed of a mother and her baby playing, and are rated from 0-14 for aspects of maternal behaviour, aspects of infant behaviour, and dyadic synchrony, whereby a higher score indicates greater amounts of that behaviour present.
Time Frame: Compare changes between baseline and week 6
Reporting Status: Not Posted

8. Secondary Outcome: To Ascertain Whether Online Singing Improves the Perceived Mother-infant Relationship Using the Maternal Postpartum Attachment Scale (MPAS)
Description: To assess whether the online singing intervention improves upon aspects of the mother-infant relationship.
  The perceived mother-infant relationship will be assessed using:
  Maternal Postpartum Attachment Scale (MPAS): The MPAS is a 19-item questionnaire assessing maternal feelings of attachment and bonding towards her baby. Items are rated from 1 to 5, whereby a lower score indicates less bonding/attachment with her baby.
Time Frame: Compare changes between baseline and weeks 6 and 32.
Reporting Status: Not Posted

9. Secondary Outcome: To Ascertain Whether Online Singing Improves the Perceived Mother-infant Relationship Using the Parent Reflective Functioning Questionnaire (PRFQ)
Description: To assess whether the online singing intervention improves upon aspects of the mother-infant relationship.
  The perceived mother-infant relationship will be assessed using:
  Parent Reflective Functioning Questionnaire (PRFQ): The PRFQ is an 18-item questionnaire that asks mothers to reflect on their relationship with their infant and how attuned they perceive themselves to be. It assesses a caregiver's capability to reflect upon her own internal mental experiences as well as those of the baby. Each item is rated on a likert scale from 1 (strongly disagree) to 7 (strongly agree) with a total possible score ranging from 18-126.
Time Frame: Compare changes between baseline and weeks 6 and 32.
Reporting Status: Not Posted

10. Secondary Outcome: To Ascertain Whether Online Singing Improves Social Support and Reduces Loneliness Using the UCLA Loneliness Scale
Description: To assess whether the online singing intervention improves aspects of loneliness and perceived support.
  UCLA Loneliness Scale: is a 20-item questionnaire that assesses one's perceived sense of loneliness. Questions address relationships and loneliness. Items are rated as 'often,' 'sometimes,' 'rarely,' or 'never.' Scores can range from 20-80, whereby a higher score indicates a greater sense of loneliness.
Time Frame: Compare changes between baseline and weeks 3, 6, 16, 32.
Reporting Status: Not Posted

11. Secondary Outcome: To Ascertain Whether Online Singing Improves Social Support and Reduces Loneliness Using the Multidimensional Scale of Perceived Social Support (MSPSS)
Description: To assess whether the online singing intervention improves aspects of loneliness and perceived support.
  Multidimensional Scale of Perceived Social Support (MSPSS): is a 12-item questionnaire that assesses perceived support (practical and emotional) from peers, family, and friends. Each item is rated from 1 (very strongly disagree) to 7 (very strongly agree) and is scored from 12-84, where a higher score indicates a greater sense of perceived social support.
Time Frame: Compare changes between baseline and weeks 3, 6, 16, 32.
Reporting Status: Not Posted

12. Secondary Outcome: To Identify Whether There Are Biological Mechanisms Underpinning the Psychological Outcomes Assessed Using Changes in Measurements in Stress Hormones, Including Diurnal Cortisol and Salivary Cytokines
Description: Stress hormones, including diurnal cortisol and salivary cytokines. These measures will be analysed using an array of techniques including enzyme-linked immunosorbent assay (ELISA). Higher levels of cortisol and cytokines may indicate higher levels of stress.
Time Frame: Compare changes between baseline and week 6 (end of treatment).
Reporting Status: Not Posted

13. Secondary Outcome: To Identify Whether There Are Biological Mechanisms Underpinning the Psychological Outcomes Assessed Using Changes in Measurements in Salivary Oxytocin
Description: Levels of salivary oxytocin measured. These measures will be analysed using an array of techniques including enzyme-linked immunosorbent assay (ELISA). Higher levels of oxytocin may indicate positive interactions between mothers and babies.
Time Frame: Compare changes between baseline and week 6 (end of treatment).
Reporting Status: Not Posted

14. Secondary Outcome: To Identify How the Online Singing Sessions Affect the Lived Experience of Mothers With PND Using Focus Groups
Description: Focus groups: focus groups will take place immediately following session 6 (if logistically possible) for all mothers focusing on their lived experience of the intervention and their reported mechanisms of effect
Time Frame: Qualitative data collection at week 6 (end of intervention).
Reporting Status: Not Posted

15. Secondary Outcome: To Explore the Phenomenology of PND and How Singing Intersects With PND Among Women With Particular Risk Factors for PND (Traumatic Birth, Adverse Childhood Experiences, and Social Isolation/Loneliness) Using Semi-structured Interviews
Description: Semi structured interviews: individual or small-group interviews with three sub-groups of women self-reporting particular risk factors for PND: traumatic birth, adverse childhood experiences, and social isolation/loneliness. These interviews will focus in-depth on the phenomenology of PND and how singing intersects with the specific context of PND among the sub-groups.
Time Frame: Qualitative data collection at week 6 (end of intervention).
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 months.
Arm/Group | M4M Intervention
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT04857593/Prot_SAP_000.pdf